CLINICAL TRIAL: NCT06478550
Title: A Pilot Study Investigating the Effect of Patient Support Solution App With Connectivity on Once-weekly Semaglutide s.c. Treatment Persistence in Patients With Type 2 Diabetes in a Clinical Practice Setting
Brief Title: A Research Study to Understand How People With Type 2 Diabetes Take Ozempic® and if the Ozempic®App Helps Them Stay on This Treatment
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-5029; U1111-1286-4221 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient Support Solution (PSS) app with connectivity to Mallya: Participants will be treated with commercially available semaglutide subcutaneously (s.c.) according to routine clinical practice and local label at the discretion of the Health Care Providers (HCP) and receive PSS app with connectivity to Mallya device.
  Interventions: Drug: Semaglutide
- PSS app without connectivity to Mallya: Participants will be treated with commercially available semaglutide s.c. according to routine clinical practice and local label at the discretion of the HCP and receive PSS app without connectivity to Mallya device.
  Interventions: Drug: Semaglutide
- Mallya: Participants will be treated with commercially available semaglutide s.c. according to routine clinical practice and local label at the discretion of the HCP and use only Mallya device without PSS app.
  Interventions: Drug: Semaglutide
- No intervention (Control arm): Participants will be treated with commercially available semaglutide s.c. according to routine clinical practice and local label at the discretion of the HCP and will not receive PSS app or Mallya device.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will be treated with commercially available semaglutide subcutaneously (s.c.) according to routine clinical practice and according to local label at the discretion of the Health Care Providers (HCP). The decision to initiate treatment with semaglutide s.c. is independent from the decision to include the participant in the study.
  Other Names: Ozempic®

SUMMARY:
This study looks at how participants with type 2 diabetes take Ozempic® and if the Ozempic® app helps participants to stay on this treatment. Participants will already be prescribed with Ozempic® by the study doctor. Participants may be asked to use a device called Mallya®, which participants must attach to their Ozempic® injection pen. Participants might also be asked to install an Ozempic® app on their mobile phone which supports the participants in the use of Ozempic®. At the beginning and at the end of this study, the participants will have to fill out some questionnaires about their diabetes treatment. Participants may also be chosen to participate in a voluntary non-mandatory interview after the study has ended. The total duration of study is approximately 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available semaglutide s.c. has been made by the patient and the Health Care Providers (HCP) and independently from the decision to include the patient in this study. Patients can be randomised up to 10 days after being prescribed semaglutide.
* Treatment with semaglutide s.c. is needed for intensification of glycaemic control and used according to label as judged by HCP.
* Male or female; aged 25-75 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 2 diabetes (T2D) at least 180 days prior to obtaining informed consent.
* Willing to comply with the protocol requirements which includes use of Patient Support Solution (PSS) app on own mobile device (iphone Operating System (iOS) 11 (or higher) and Android 4.1 (or higher) devices), using Mallya®, filling out questionnaires as judged by the HCP.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Glucagon Like Peptide-1 Receptor Agonist (GLP-1 RA) use for 90 days prior to randomisation. However, one prescription of once-weekly semaglutide subcutaneously (s.c.) is allowed up to 10 days prior to randomisation.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Use of pacemaker or body worn infusion pumps according to Mallya®'s instruction for use.
* Impaired eyesight prohibiting readability of PSS app provided on mobile device.
* Inability to independently self-manage anti-diabetic treatments received as judged by HCP.
* Inability to independently inject semaglutide s.c. treatment as judged by HCP.
* Inability to fulfil study requirement as judged by the HCP.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Persistency of semaglutide s.c. treatment in PSS app with connectivity vs control arm (Yes/No) (HCP reported) | At Visit 2 (week 16)
  Measured as number of participants (Yes/No).

SECONDARY OUTCOMES:
Time from first dose to discontinuation (HCP reported) | From Visit 1 (week 0) to Visit 2 (week 16)
  Measured in days.
HCP prespecified maintenance dose achieved at V2 (week 16) | At visit 2 (week 16)
  Measured as number of participants (Yes/No).
Time to HCP prespecified maintenance dose (HCP reported) | From Visit 1 (week 0) to Visit 2 (week 16)
  Measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (6):
- Greece (6):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki, Nea Efkarpia
  - "Laiko" General Hospital of Athens, Goudi/Athens
  - Univ Gen Hospital Larisa, Larissa
  - Geniko Nosokomeio Peiraia Tzaneio, Piraeus
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com